CLINICAL TRIAL: NCT03283267
Title: A Single-center Safety and Pharmacodynamic Study of Healthy Chinese Subjects Administered Sodium Zirconium Cyclosilicate (ZS)
Brief Title: A Safety and Pharmacodynamic Study of Healthy Chinese Subjects Administered Sodium Zirconium Cyclosilicate (ZS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9483C00001
Record Dates: First submitted 2017-08-21; First posted 2017-09-14 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Hyperkalemia
Keywords: Healthy Chinese Subjects, Pharmacodynamic Study
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZS 5g, qd (Experimental): Subjects randomized to this arm will receive ZS 5 g qd in conjunction with breakfast during the ZS treatment period and will be continued with a standard diet.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS)
- ZS 10g, qd (Experimental): Subjects randomized to this arm will receive ZS 10 g qd in conjunction with breakfast during the ZS treatment period and will be continued with a standard diet.
  Interventions: Drug: Sodium Zirconium Cyclosilicate (ZS)

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (ZS) — Sodium zirconium cyclosilicate (ZS) is a non-absorbed, inorganic crystalline compound that selectively captures potassium ions in exchange for sodium and hydrogen ions in the gastrointestinal tract after oral administration.

SUMMARY:
This is a single center, inpatient, open label pharmacodynamic study to determine the effect of 5 g and 10 g doses of Sodium Zirconium Cyclosilicate (ZS) administered once daily (qd) for 4 days on potassium and sodium excretion in healthy Chinese subjects on a standardized, low sodium and high potassium diet.

DETAILED DESCRIPTION:
This study will be conducted at 1 study centre in Hong Kong. Approximately 22 Subjects will be screened to achieve 20 subjects completing the study. Subjects will be randomized to receive ZS 5 g or 10 g (1:1) once daily (qd) in conjunction with breakfast and will be continued with a standard diet during the ZS treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and/or male healthy Chinese subjects aged between 18 and 55 inclusive who reside in Hong Kong
3. Ability to have repeated blood draws or effective venous catheterization
4. Willing to consume food and beverages using a standardized daily diet containing 40 (± 10%) mEq/day sodium and 128 (± 10%) mEq/day potassium provided by the research site

Key Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 months
2. Subjects who were receiving concomitant medications including vitamins, dietary supplements and herbal preparations within 2 weeks prior to Study Day 1 of the Diet Run-in Period.
3. Current and/or past history of alcohol abuse within the past year or a positive results (exceed normal range) of breath test for alcohol abuse
4. Current and/or past history of drugs abuse within the past year or a positive drug abuse screen, e. g. methylenedioxymethamphetamine, opiate, barbiturates, benzodiazepines, ketamine, cocaine, amphetamine, methamphetamine, marijuana, and methadone.
5. Plasma donation within 1 month of screening or any blood donation/blood loss >500 mL during the 3 months prior to screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to ZS treatment period in urine potassium excretion. | Study Day 3 and 4 vs Study Day 7 and 8.
  The 48- hour urine potassium excretion on Study Days 3 and 4 (baseline) will be compared with 48-hour urine potassium excretion on Study Days 7 and 8 (on study drug).

SECONDARY OUTCOMES:
Mean change from baseline to ZS treatment period in urine sodium excretion. | Study Day 3 and 4 vs Study Day 7 and 8.
  The 48- hour urine sodium excretion on Study Days 3 and 4 (baseline) will be compared with 48- hour urine sodium excretion on Study Days 7 and 8 (on study drug).
Mean change from baseline to ZS treatment period in serum potassium (S-K). | Study Day 3 and 4 vs Study Day 7 and 8.
  Mean change in S-K from the Baseline Period (Day 3 and 4) to the ZS Treatment Period (Day 7 and 8).

OTHER OUTCOMES:
Number of subjects with adverse events | From Day 1 through Follow-up visit
Changes in vital signs | Through study completion, up to 10 days
Changes in standard Electrocardiograph (ECG ) parameters | Through study completion, up to 10 days
Changes in standard physical examination parameters including height | Through study completion, up to 10 days
Changes in standard clinical chemistry lab parameters | Through study completion, up to 10 days
Changes in standard hematology lab parameters | Through study completion, up to 10 days
Changes in Serum calcium (S-Ca) | Through study completion, up to 10 days
Changes in Serum magnesium (S-Mg) | Through study completion, up to 10 days
Changes in Serum sodium (S-Na) | Through study completion, up to 10 days
Changes in Serum phosphate (S-PO4) | Through study completion, up to 10 days
Changes in Serum bicarbonate (S-HCO3) | Through study completion, up to 10 days
Changes in Blood urea nitrogen (BUN) | Through study completion, up to 10 days
Number of subjects with Serious adverse events | Through study completion and follow-up visit, up to 34 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No